CLINICAL TRIAL: NCT01233167
Title: Benefits and Risks Evaluation of Different Anti-platelet Strategies Beyond a 12-month Period Inpatients Receiving Sirolimus Drug-eluting Stent Implantation
Brief Title: Effect of Different Anti-platelet Strategies on the Long-term Outcome After Sirolimus Drug-eluting Stent Implantation
Acronym: EASTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Guosheng Fu, director of cardiovascular department, Sir Run Run Shaw Hospital, College of medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SRRSH-CVD-001
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Artery Disease
Keywords: dual antiplatelet therapy; sirolimus drug-eluting stent; major adverse cardiac events; bleeding
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Hemorrhage | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- clopidogrel (Experimental)
  Interventions: Drug: clopidogrel
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- steply discontinued clopidogrel (Experimental)
  Interventions: Drug: clopidogrel and placebo

INTERVENTIONS:
Drug: clopidogrel — clopidogrel 75 mg po per day for 12 months
  Arms: clopidogrel
Drug: placebo — placebo 75mg po per day for 12 months
  Arms: placebo
Drug: clopidogrel and placebo — clopidogrel 50mg per day for 3 months,clopidogrel 25mg per day for 3 months,then placebo 75mg per day for 6 months
  Arms: steply discontinued clopidogrel

SUMMARY:
The study aims to assess the effectiveness of dual antiplatelet therapy, aspirin alone versus steeply discontinued clopidogrel plus aspirin in preventing clinical MACE events.Our subject is beyond a 12-month period patients receiving sirolimus drug-eluting stent implantation.

DETAILED DESCRIPTION:
It is not clear that dual antiplatelet therapy is better than aspirin beyond 12-months period patients receiving sirolimus drug-eluting stent implantation. If aspirin plus clopidogrel reduced MACE rates without increasing blood events, the investigators will evaluate risk-benefit ratio. The investigators will observe all cause mortality, nonfatal myocardial infarction, or clinical-driven target vessel revascularization TVR in a 1-year trial duration. In addition, strokes, stent thrombosis, cardiac re-hospitalizations, dialysis/hemofiltration, duration of hospitalization and bleeding events will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of older.
* The latest PCI with DES implantation before 12 months (stents must be one or more sirolimus-eluting stents).
* Angiographically confirmed major epicardial vessels (>=2.5mm in diameter) without significant stenosis or restenosis (>=50%).
* Geographically accessible and willing to come in for required study visits.
* Signed informed consent.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to aspirin and clopidogrel.
* Severe congestive heart failure (class III or IV according to NYHA, or pulmonary edema) at the time of enrollment and within 12 months.
* EF<35% within 12 months.
* Severe cardiac valves disease, or idiopathic cardiomyopathy such as dilated cardiomyopathy, hypotrophic cardiomyopathy. Other severe system diseases.
* Previous ACS within 12 months.
* Previous stroke or transient ischemia attack within 12 months.
* Previous myocardial infarction and clinical-driven target vessel revascularization within 12 months.
* Current enrollment in another clinical trial.
* Suspected pregnancy.
* Big bleeding events within 12 months.
* Planned surgical procedure.
* Previous other type DES implantation or BMS implantation history.
* Extra-cardiac stent implantation history.
* Current or planned dialysis.
* The patient has a known hypersensitivity or contraindication to statins.
* Current or planned high dose and long-term glucocorticoid treatment.
* that is expected to limit survival to less than 1 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5232 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year
nonfatal myocardial infarction | one year
clinical-driven target vessel revascularization | one year
cardiac death | one year
stent thrombosis | one year

SECONDARY OUTCOMES:
death | one year
myocardial infarction | one year
any repeat revascularization | one year
strokes | one year
dialysis/hemofiltration | one year
bleeding events | one year